CLINICAL TRIAL: NCT02426268
Title: CAS Medical Systems FORE-SIGHT Elite Tissue Oximeter During Cardiac Surgery
Brief Title: FORE-SIGHT Tissue Oximeter During Cardiac Surgery
Acronym: FORE-SIGHT
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: CAS Medical Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Emily Methangkool, MD, MPH, Assistant Clinical Professor, University of California, Los Angeles
Other Study IDs: FORE-SIGHT 13-000448
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Surgical Patients
Keywords: cardiac surgery; cerebral oximetry; lower extremity oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to measure cerebral and lower extremity oximetry on patients during cardiac surgery.

DETAILED DESCRIPTION:
The purpose of this research study is to collect data from a tissue oximeter device that measures brain oxygen saturation simultaneous with data from the same device that monitors skeletal muscle during cardiac surgery. This monitoring will allow for continuous, non-invasive, and earlier assessment of perfusion abnormalities/hypoperfusion.

Two sensors from the FORE-SIGHT Elite monitor will be placed on the forehead above the eyebrows and two additional sensors will be placed on the leg muscles. Data from the FORE-SIGHT Elite monitor will be recorded in addition to clinical and demographic data, which is standard of care during the procedure, for research purposes to look at factors associated with desaturations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects where cerebral oximetry is monitored during their surgery

Exclusion Criteria:

* Birthmarks, tattoos, or other skin abnormalities that FORE-SIGHT Sensors cannot avoid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiothoracic surgical population at UCLA
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Cerebral Oxygen Saturation | Duration of the surgery (~5-7 hours)
  Two sensors from FORE-SIGHT Elite monitor will be placed on the forehead above the eyebrows to continuously monitor cerebral oxygen saturation.

SECONDARY OUTCOMES:
Non-Cerebral Oxygen Saturation | Duration of the surgery (~5-7 hours)
  Two sensors from FORE-SIGHT Elite monitor will be placed on the leg muscles to continuously monitor non-cerebral/skeletal muscle oxygen saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Methangkool, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology, Los Angeles, California, United States